CLINICAL TRIAL: NCT06806956
Title: Severe Malaria Treatment With Rectal Artesunate and Artemisinin-based Combination Therapy in Remote Settings
Brief Title: Severe Malaria in Remote Areas- Closing the Evidence Gap
Acronym: SEMA ReACT
Status: Enrolling by invitation | Type: Observational
Sponsor: Tropical Diseases Research Centre, Zambia (Other Government)
Collaborators: Universiteit Antwerpen (Other); University of Kinshasa (Other); National Institute for Medical Research, Tanzania (Other Government); Medicines for Malaria Venture (Other); Université de Lubumbashi (Other)
Responsible Party: Sponsor
Other Study IDs: Version 2.0 Dated 5 March 2024; 101103191 (Other Grant/Funding Number: HORIZON-JU-GH-EDCTP3-2022-CALL1-01-01)
Record Dates: First submitted 2024-11-29; First posted 2025-02-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Severe Malaria
Keywords: Rectal artesunate; Artemisinin-based Combination Therapy; Injectable artesunate; Community Health Worker; Health Facility
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We are collecting Dried Blood Spots for looking at markers of resistance for malaria
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Two groups i.e rectal artesunate +ACT group while the other is injectable artesunate +ACT group: The group of interest is children aged between 6 months and less than or equal to 5 years with severe malaria. However, we will also enrol children of the same age group with simple malaria and non malaria severe disease to compare their journeys as well
  Interventions: Drug: Treatment of severe malaria with either RAS + ACT or RAS + injectable artesunate + ACT will each achieve the clinically acceptable cure rate of 97% ± 5% in remote areas

INTERVENTIONS:
Drug: Treatment of severe malaria with either RAS + ACT or RAS + injectable artesunate + ACT will each achieve the clinically acceptable cure rate of 97% ± 5% in remote areas — The Community Health Worker will give rectal artesunate (RAS) +artemisinin based combination Therapy (ACT) to children aged 6 months to less than or equal to 5 years who fail to make the referral trip. Those who make the referral trip will receive injectable artesunate and artemisinin based Combination Therapy for three days. Giving of RAS +ACT is unique to this study. Children with non malaria severe disease will also receive amoxicillin from the community health worker before they are referred to the next level of care

SUMMARY:
The goal of this observational study is to assess whether the giving of rectal artesunate and a three day course of an Artemisinin based Combination Therapy (ACT) to children aged 6 months and ≤ 5 years with severe malaria when referral is not feasible is non inferior to giving of injectable artesunate and three day course of an ACT. The three primary objectives are:

* To evaluate the 28-day PCR corrected cure rate in children aged 6 months to ≤ 5 years treated with RAS+ACT or RAS+injectable artesunate, assessing whether each treatment achieves the clinically acceptable cure rate of 97% ± 5%.
* To evaluate feasibility of provision of rapid treatment of severe malaria with rectal artesunate in children 6 months to ≤ 5 years not able to access a referral health facility, by a community health worker or in health facility where there is no injectable artesunate available.
* To evaluate the impact of reinforcing the integrated Community Case Management (iCCM) on access to the formal health care system

The study is being done in Nchelenge district in Zambia and Kapolowe district in the Democratic Republic of Congo. It will enrol 1008 children with severe malaria and an equal number of children with simple malaria

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for severe malaria

* From a village without other research interventions
* Children aged from 6 months to ≤5 years that present at the health system and are either; with fever (or history of fever within 2 days) and have a positive mRDT test plus at least one of the following danger signs for malaria (as per standardized national iCCM guidelines):

  * convulsions
  * inability to drink, eat, or suck
  * vomiting all liquids and solids
  * altered consciousness/coma
  * lethargy
  * chest in-drawing Inclusion for uncomplicated malaria
* Children aged from 6 months to ≤5 years; with fever (or history of fever within 2 days) with no danger signs for malaria (as per the standardized national Integrated Management of Childhood Illnesses guidelines) with a positive mRDT for Plasmodium falciparum histidine-rich protein.

Inclusion for severe non-malaria

* From a village without other research interventions
* Children aged from 6 months to ≤5 years that present at the health system and are either; with fever (or history of fever within 2 days) and have a negative mRDT test plus at least one of the following danger signs as per standardized national iCCM guidelines:

  * convulsions
  * inability to drink, eat, or suck
  * vomiting all liquids and solids
  * altered consciousness/coma
  * lethargy
  * chest in-drawing
* For participants in sentinel sites, a written informed consent will be provided by the patient's parent or guardian to take filter paper blood samples and to participate in interviews (questionnaires and IDI) at enrolment, day 14 and day 28 (to assess malaria recurrence and look for markers of resistance). If the parent or guardian is unable to write, thumb print witnessed consent is permitted. The informed consent shall be administered by the CHWs. Willingness and ability of the patient and the parent or guardian to comply with the treatment policy.

Exclusion Criteria:

* Use of any investigational or non-registered product or planned use during the study period.
* Participation in other studies within 30 days before the current study begins and/or during study participation.
* Inability to comprehend and/or unwillingness to follow the study protocol.
* For RAS use: if the child has reacted badly to artesunate in the past (in sites where RAS is administered)

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will comprise children 6 months to ≤5 years of age living in Kapolowe, DRC and those living in Nchelenge, Zambia who present with a suspected diagnosis of severe malaria or uncomplicated malaria, confirmed by a rapid diagnostic test; or non-malaria severe disease
Sampling Method: Non-Probability Sample
Enrollment: 2016 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
The time from onset of symptoms to initiating treatment | The time from onset of symptoms to initiating treatment
  The time from onset of symptoms to initiating treatment among children 6 months to ≤5 years with severe malaria and/or not able to take oral treatment that seek health care from the CHW or other HF system as primary first contact
PCR-corrected cure rate at 28 days from enrollment in patients aged 6 months to ≤5 years. | 28 Days from enrollment
  PCR-corrected cure rate at 28 Days from enrollment in patients aged 6 months to ≤5 years in areas where referral for follow-up treatment with injectable artesunate is not feasible, compared to outcomes obtained after full referral is completed
Change from baseline proportion of sick children 6 months - ≤5 years at population level that went to the formal health system during the last 6 months including suspected (severe) malaria at month 20 (phase 4). | At month 20 (phase 4)
  Two cross section surveys one at month 1 (baseline) and the other at month 20 (phase 4) will be used to obtain the proportion of sick children 6 months to ≤5 years at population level that were either attended by a Community Health Worker, Health post or Health Centre in the last 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- University of Kinshasa, Kinshasa, Kinshasa City, Democratic Republic of the Congo
- Tropical Diseases Research Centre, Ndola, Copperbelt, Zambia

IPD SHARING:
Plan to Share IPD: No
We will only share aggregated data as IPD will not be useful to the research community